CLINICAL TRIAL: NCT07184580
Title: Electrical Impendance Tomography Usage in ICU : Registry Creation
Brief Title: Electrical Impendance Tomography Usage in ICU
Acronym: EITICU
Status: Not yet recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Charles Dehout, Medical doctor, intensivist, principal investigator, Erasme University Hospital
Other Study IDs: HUB2025218
Record Dates: First submitted 2025-08-26; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: ARDS; Alveolar Recruitment Manoeuvres; Prone Position; Electrical Impedance Tomography (EIT)
Keywords: ARDS; Recruitment manoeuvres; Prone positioning; PEEP optimization; EIT; Electrical impedance tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mechanically ventilated patients: Mechanically ventilated patients for which an EIT belt has been placed, for PEEP optimization, ventilation monitoring, prone positioning evaluation,...
- Non-invasive ventilation patients: Patients included in the study who are only on

SUMMARY:
Electrical Impedance Tomography (EIT) is a non-invasive, radiation-free, bedside imaging technique that has been in clinical use for over three decades (1).

It is primarily utilized to monitor regional lung ventilation in mechanically ventilated patients. In recent years, EIT has become a routine tool in critical care settings due to its capacity to provide real-time, bedside insights into pulmonary function. Its applications are diverse, ranging from support during non-invasive ventilation and endotracheal intubation (2) to the management of complex cases of mechanical ventilation. One of its key advantages lies in guiding the optimization of Positive End-Expiratory Pressure (PEEP) titration, which may help tailor ventilatory support to individual patients and potentially reduce the mechanical power delivered to the lungs(3,4).

Despite these benefits, current evidence does not conclusively demonstrate a reduction in mortality associated with the use of EIT in critical care (5,6). Nevertheless, EIT shows promise in several emerging areas, such as monitoring ventilation distribution during prone positioning - even in awake, non-intubated patients (7) - and in the early detection of atelectasis under various clinical conditions (8).

Recently, advancements in EIT technology have led to the development of new models capable of assessing pulmonary "pulsatility," thereby expanding the potential clinical applications of EIT beyond traditional ventilation monitoring. This feature may facilitate the bedside detection of conditions such as atelectasis, pneumonia, pleural effusion, and even pulmonary embolism (9,10).

In this context, the Intensive Care Unit at Erasme Hospital is acquiring two EIT devices to enhance diagnostic capabilities and improve the care of patients requiring either non-invasive or invasive ventilation during their ICU stay. To support the systematic implementation of these devices and enable future research, it is necessary to establish a registry documenting their clinical use within the ICU. This registry will serve as a foundation for tracking usage patterns, evaluating outcomes, and potentially contributing to future scientific studies.

Standard ICU data such as SOFA scores and SAPS II will be recorded, as is already routinely done in some registries like Epimed.

This registry will be specific to the Erasme ICU and will collect detailed data on ventilation parameters, EIT measurements, and recruitment maneuvers in patients undergoing mechanical ventilation-whether invasive or non-invasive-when the clinical team determines that a recruitment maneuver is indicated and chooses to use an EIT device for monitoring.

Data will be entered into RedCap by the attending physicians or physiotherapists responsible for the patient.

Data collection will be prospective, as it is not technically possible to automatically synchronize the recording of ventilation parameters and EIT measurements using the existing software systems.

There are no expected risks for the patients, as the procedures involved are considered standard practice in intensive care settings.

Patients may benefit from the collection of these data, as it allows for closer monitoring of ventilation parameters during their ICU stay.

As this is a registry-based study, there will be no predefined duration or fixed number of patients. However, we estimate data will be recorded over a five-year period, with an inclusion of at least 300 patients per year.

Inclusion Criteria for ICU Patients:

* Patient aged more than 12 years old (no pediatric EIT belt)
* Patient monitored by an EIT belt OR Patient undergoing a recruitment maneuver OR Patient undergoing prone position.

ELIGIBILITY:
Inclusion Criteria for ICU Patients:

* Patient aged more than 12 years old (no pediatric EIT belt)
* Patient monitored by an EIT belt

Exclusion criteria Patient who expressed opposition to participate.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All critical care patients for whom clinicians estimated the need for EIT measurements could be included, except pediatric patients under 12 years of age, as the belt used for this device is not designed for children.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | up to 30 days
  Assessment of mortality

SECONDARY OUTCOMES:
PaO2/FiO2 ratio | During the measurement using the EIT in the ICU
  Measurement on PaO2/FiO2 before and after the usage of EIT
Hospital mortality rate | Through hospital discharge (average of 14 days)
  Hospital mortality
Ventilation free days | 28 days since the start of ventilation
  Number of days without ventilation for patients who are mechanically ventilated
Mechanical power | During the measurement using the EIT in the ICU
  Measurement on mechanical power before and after the usage of EIT

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beitler JR, Sarge T, Banner-Goodspeed VM, Gong MN, Cook D, Novack V, Loring SH, Talmor D; EPVent-2 Study Group. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):846-857. doi: 10.1001/jama.2019.0555. PMID 30776290
- [Background] He H, Chi Y, Yang Y, Yuan S, Long Y, Zhao P, Frerichs I, Fu F, Moller K, Zhao Z. Early individualized positive end-expiratory pressure guided by electrical impedance tomography in acute respiratory distress syndrome: a randomized controlled clinical trial. Crit Care. 2021 Jun 30;25(1):230. doi: 10.1186/s13054-021-03645-y. PMID 34193224
- [Background] Songsangvorn N, Xu Y, Lu C, Rotstein O, Brochard L, Slutsky AS, Burns KEA, Zhang H. Electrical impedance tomography-guided positive end-expiratory pressure titration in ARDS: a systematic review and meta-analysis. Intensive Care Med. 2024 May;50(5):617-631. doi: 10.1007/s00134-024-07362-2. Epub 2024 Mar 21. PMID 38512400
- [Background] Jimenez JV, Munroe E, Weirauch AJ, Fiorino K, Culter CA, Nelson K, Labaki WW, Choi PJ, Co I, Standiford TJ, Prescott HC, Hyzy RC. Electric impedance tomography-guided PEEP titration reduces mechanical power in ARDS: a randomized crossover pilot trial. Crit Care. 2023 Jan 17;27(1):21. doi: 10.1186/s13054-023-04315-x. PMID 36650593
- [Background] Kim Y, Webster JG, Tompkins WJ. Electrical impedance imaging of the thorax. J Microw Power. 1983 Sep;18(3):245-57. doi: 10.1080/16070658.1983.11689329. PMID 6558130